CLINICAL TRIAL: NCT05842460
Title: Testing the Impact of an "Ultraprocessed" Front-of-package Warning Label Among Brazilian Consumers
Brief Title: Testing "Ultraprocessed" Front-of-package Label Among Brazilian Consumers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Bloomberg Family Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-0151
Record Dates: First submitted 2023-03-15; First posted 2023-05-06 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Dietary Exposure
MeSH Terms: interventions — Nutrients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrient warnings (Active Comparator): Individuals in this trial arm will see images of products carrying nutrient warnings that are currently included in Brazil's front-of-package labeling scheme.
  Interventions: Behavioral: Nutrient warning labels
- Nutrient and ultraprocessed warnings (Experimental): Individuals in this trial arm will see images of products carrying nutrient warnings that are currently included in Brazil's front-of-package labeling scheme and an experimental warning stating that the product is ultraprocessed.
  Interventions: Behavioral: Nutrient and ultraprocessed warning labels

INTERVENTIONS:
Behavioral: Nutrient warning labels — Inclusion of nutrient warning labels, which are currently mandatory in Brazil, to images of food products.
  Arms: Nutrient warnings
Behavioral: Nutrient and ultraprocessed warning labels — Inclusion of nutrient warning labels, which are currently mandatory in Brazil, and an experimental ultraprocessed warning label to images of food products.
  Arms: Nutrient and ultraprocessed warnings

SUMMARY:
The goal of this experiment is to test the effects an "ultraprocessed" warning label on foods and beverages among Brazilian consumers. The main questions it aims to answer are:

* Do "ultraprocessed" warnings affect Brazilian consumers' intention to purchase products?
* Do "ultraprocessed" warnings affect Brazilian consumers' product perceptions?

Participants will see images of four products carrying either nutrient warning labels (which are currently mandatory in Brazil) or nutrient warning labels alongside an experimental warning label informing that the product is ultraprocessed. Participants will then answer survey questions about each product. Researchers will compare responses between both arms to determine if the "ultraprocessed" warning significantly changes the effect of nutrient warnings.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older,
* residing in Brazil,
* responsible for at least 50% of the household's grocery purchases.

Exclusion criteria:

* involvement in any pre-testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Purchase intentions | Online survey within 20 minutes following completion of a ~10 minute shopping task.
  How likely the participant would be to buy products will be measured by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher likelihood of buying products.

SECONDARY OUTCOMES:
Product healthfulness perceptions | Online survey within 20 minutes following completion of a ~10 minute shopping task.
  How healthy products seem to the participant will be measured by survey. Response options are on a 1 to 5 scale, with higher scores representing a higher perceived product healthfulness.
Product processing status perceptions | Online survey within 20 minutes following completion of a ~10 minute shopping task.
  Whether the participant believes products are ultraprocessed will be measured by survey. Responses options are "no," "yes," and "I'm not sure."
Message effectiveness perceptions | Online survey within 20 minutes following completion of a ~10 minute shopping task.
  Perceived message effectiveness of the study labels will be measured by survey through a three-item scale. Items inquire about how much the labels discourage the participant from wanting to consume the products, how much the labels make the participant concerned about the health effects of consuming the products, and how much the labels make consuming the products seem unpleasant. Response options are on a 1 to 5 scale, with higher scores representing a higher perceived message effectiveness of the study labels.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset and analytic code will be uploaded to a public repository upon publication of the study.
Supporting Information: Analytic Code
Time Frame: Upon publication of the study.
Access Criteria: No access criteria. The dataset and analytic code will be made publicly available at Open Science Framework.

REFERENCES:
- [Background] Cotter T, Kotov A, Wang S, Murukutla N. 'Warning: ultra-processed' - A call for warnings on foods that aren't really foods. BMJ Glob Health. 2021 Dec;6(12):e007240. doi: 10.1136/bmjgh-2021-007240. No abstract available. PMID 34933866
- [Background] Romero Ferreiro C, Lora Pablos D, Gomez de la Camara A. Two Dimensions of Nutritional Value: Nutri-Score and NOVA. Nutrients. 2021 Aug 13;13(8):2783. doi: 10.3390/nu13082783. PMID 34444941
- [Derived] D'Angelo Campos A, Ng SW, Duran AC, Khandpur N, Taillie LS, Christon FO, Hall MG. "Warning: ultra-processed": an online experiment examining the impact of ultra-processed warning labels on consumers' product perceptions and behavioral intentions. Int J Behav Nutr Phys Act. 2024 Oct 9;21(1):115. doi: 10.1186/s12966-024-01664-w. PMID 39385224
- See also: Related Info — https://www.medrxiv.org/content/10.1101/2022.11.18.22282494v1

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT05842460/SAP_000.pdf